CLINICAL TRIAL: NCT05459233
Title: Valve Hemodynamic Optimization Based on Doppler-Echocardiography Versus Catheterization Measurements Following Valve-in-Valve TAVR: A Prospective Randomized Trial
Brief Title: Valve Hemodynamic Optimization Based on Doppler-Echocardiography vs Catheterization Measurements Following ViV TAVR
Acronym: ECHOCATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECHOCATH
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Regurgitation; Prosthesis Failure
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion to valve hemodynamic optimization according to Doppler-echocardiography versus cardiac catheterization parameters.
Who Masked: Participant
Masking Description: Single-blinded trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doppler-echocardiography (Other): Following valve implantation, further intervention will be based on Doppler-echocardiographic measurements.
  Interventions: Procedure: Doppler-echocardiography
- Invasive hemodynamic measurements (Other): Following valve implantation, further interventions will be based on invasive hemodynamic measurements (with simultaneous aortic and ventricular pressure recording).
  Interventions: Procedure: Invasive hemodynamic measurements

INTERVENTIONS:
Procedure: Doppler-echocardiography — The TAVR (valve-in-valve) procedure will be performed with the SAPIEN 3 Ultra valve, with valve sizing according to current manufacturer recommendations. Following valve implantation, further intervention will be based on Doppler-echocardiographic measurements. Balloon post-dilation with a non-compliant balloon will be performed in the presence of a residual mean gradient ≥20 mmHg as assessed by Doppler-echocardiography.
  Arms: Doppler-echocardiography
Procedure: Invasive hemodynamic measurements — The TAVR (valve-in-valve) procedure will be performed with the SAPIEN 3 Ultra valve, with valve sizing according to current manufacturer recommendations. Following valve implantation, further interventions will be based on invasive hemodynamic measurements (with simultaneous aortic and ventricular pressure recording). Balloon post-dilation will be performed with a non-compliant balloon in the presence of a mean residual gradient ≥20 mmHg as assessed by hemodynamic measurements.
  Arms: Invasive hemodynamic measurements

SUMMARY:
Data on valve performance following ViV-TAVR has usually been obtained with the use of Doppler-echocardiography. However, some reports have shown significant discordances in the evaluation of mean transvalvular gradient between echocardiography and catheterization, with an overestimation of the real gradient with echo (vs. cath) in most cases. Thus, the incidence of procedural-device failure may be lower than that reported in the ViV-TAVR literature,

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, single-blinded design trial including patients with surgical aortic bioprosthetic dysfunction in the presence of a stented surgical bioprosthesis with a labeled size ≤25 mm. Following the Heart Team's decision to proceed with a ViV-TAVR procedure with the SAPIEN 3 ULTRA valve (or its subsequent iterations), patients will be randomized to valve hemodynamic optimization according to Doppler-echocardiography versus cardiac catheterization parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical aortic bioprosthetic valve failure defined as severe aortic stenosis and/or regurgitation approved for a valve-in-valve procedure by the Heart Team
* Surgical stented bioprosthetic valve (label size ≤25 mm)
* TAVR with the SAPIEN 3 Ultra valve

Exclusion Criteria:

* Stentless or sutureless surgical valves
* Trifecta bioprosthesis
* Hancock II bioprosthesis
* High-risk of coronary obstruction (defined either as a virtual transcatheter valve - coronary distance as evaluated by CT <4 mm or based on the criterion of the heart team responsible for the procedure).
* Impossibility to obtain written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of life (Efficacy) | 12 months follow-up
  Change in quality of life as evaluated by the Kansas City Cardiomyopathy Questionnaire (KCCQ). All score are represented on a 0-to-100-point scale (lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life).The KCCQ is a 7 domains questionnaire; symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life and self-efficacy.
Periprocedural complications (Safety) | Periprocedural
  Periprocedural complications including in-hospital mortality, stroke, annular rupture, coronary obstruction, new-onset left bundle branch block, need for permanent pacemaker implantation and conversion to open heart surgery.

SECONDARY OUTCOMES:
Residual transvalvular gradient | 1 month and 12 months follow-up
  Residual (maximal and mean) transvalvular gradient
Combined enpoint: Moderate or severe prothesis-patient mismatch and/or moderate or severe aortic regurgitation (valve performance) | 1 month and 12 months follow-up
  Moderate or severe prothesis-patient mismatch (defines as an index aortic valve area 0.85-0.66 cm2/m2 (moderate), ≤0.65 cm2/m2 (severe) for patient with BMI ˂30km/m2 and 0.70-0.56 cm2/m2 (moderate), ≤0.55 cm2/m2 (severe) for patient with BMI ≥30km/m2 and/or moderate-severe aortic regurgitation (AR) (VARC-3 definition).
Heart failure | 1 and 12 months follow-up and yearly up to 5 years
  Evaluated by the New York Heart Association (NYHA) Functional Classification
Exercise capacity | 1 month and 12 months follow-up
  Exercise capacity as evaluated by the six-minute wlak test.
Changes in Quality of life | after 1-year follow-up (yearly up to 5 years)
  severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life).The KCCQ is a 7 domains questionnaire; symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life and self-efficacy.
Clinical safety endpoints | 1 and 12 months follow-up and yearly up to 5 years
  Individually and combined: death, stroke, major of lifethreatening bleeding, pacemaker implantation, myocardial infarction
re-hospitalization | 1 and 12 months follow-up and yearly up to 5 years
  Need for re-hospitalization
wear and tear deterioration (Structural valve degeneration) | 1 and 12 months follow-up and yearly up to 5 years
  wear and tear evaluated by echocardiography imaging
Leaflet disruption (Structural valve degeneration) | 1 and 12 months follow-up and yearly up to 5 years
  leaflet disruption evaluated by echocardiography imaging
flail leaflet (Structural valve degeneration) | 1 and 12 months follow-up and yearly up to 5 years
  flail leaflet evaluated by echocardiography imaging
leaflet fibrosis and/or calcification (Structural valve degeneration) | 1 and 12 months follow-up and yearly up to 5 years
  leaflet fibrosis and/or calcification evaluated by echocardiography imaging
strut fracture or deformation (Structural valve degeneration) | 1 and 12 months follow-up and yearly up to 5 years
  strut fracture or deformation evaluated by echocardiography imaging
Valve re-intervention | 1 and 12 months follow-up and yearly up to 5 years
  Need for valve re-intervention
Changes in Left ventricle mass | 1-month and 1-year follow-up
  Changes in LV mass

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (7):
- United States (6):
  - University of California, San Francisco, California
  - South Broward Hospital Disctrict D/B/A Memorial Healthcare System, Hollywood, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St-Joseph's Health INC, Syracuse, New York
  - The Christ Hospital Health Network, Cincinnati, Ohio
- IUCPQ, Québec, Quebec, Canada

REFERENCES:
- [Background] Paradis JM, Del Trigo M, Puri R, Rodes-Cabau J. Transcatheter Valve-in-Valve and Valve-in-Ring for Treating Aortic and Mitral Surgical Prosthetic Dysfunction. J Am Coll Cardiol. 2015 Nov 3;66(18):2019-2037. doi: 10.1016/j.jacc.2015.09.015. PMID 26516006
- [Background] VARC-3 WRITING COMMITTEE:; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: Updated Endpoint Definitions for Aortic Valve Clinical Research. J Am Coll Cardiol. 2021 Jun 1;77(21):2717-2746. doi: 10.1016/j.jacc.2021.02.038. Epub 2021 Apr 19. PMID 33888385
- [Background] Dvir D, Webb JG, Bleiziffer S, Pasic M, Waksman R, Kodali S, Barbanti M, Latib A, Schaefer U, Rodes-Cabau J, Treede H, Piazza N, Hildick-Smith D, Himbert D, Walther T, Hengstenberg C, Nissen H, Bekeredjian R, Presbitero P, Ferrari E, Segev A, de Weger A, Windecker S, Moat NE, Napodano M, Wilbring M, Cerillo AG, Brecker S, Tchetche D, Lefevre T, De Marco F, Fiorina C, Petronio AS, Teles RC, Testa L, Laborde JC, Leon MB, Kornowski R; Valve-in-Valve International Data Registry Investigators. Transcatheter aortic valve implantation in failed bioprosthetic surgical valves. JAMA. 2014 Jul;312(2):162-70. doi: 10.1001/jama.2014.7246. PMID 25005653
- [Background] Bleiziffer S, Simonato M, Webb JG, Rodes-Cabau J, Pibarot P, Kornowski R, Windecker S, Erlebach M, Duncan A, Seiffert M, Unbehaun A, Frerker C, Conzelmann L, Wijeysundera H, Kim WK, Montorfano M, Latib A, Tchetche D, Allali A, Abdel-Wahab M, Orvin K, Stortecky S, Nissen H, Holzamer A, Urena M, Testa L, Agrifoglio M, Whisenant B, Sathananthan J, Napodano M, Landi A, Fiorina C, Zittermann A, Veulemans V, Sinning JM, Saia F, Brecker S, Presbitero P, De Backer O, Sondergaard L, Bruschi G, Franco LN, Petronio AS, Barbanti M, Cerillo A, Spargias K, Schofer J, Cohen M, Munoz-Garcia A, Finkelstein A, Adam M, Serra V, Teles RC, Champagnac D, Iadanza A, Chodor P, Eggebrecht H, Welsh R, Caixeta A, Salizzoni S, Dager A, Auffret V, Cheema A, Ubben T, Ancona M, Rudolph T, Gummert J, Tseng E, Noble S, Bunc M, Roberts D, Kass M, Gupta A, Leon MB, Dvir D. Long-term outcomes after transcatheter aortic valve implantation in failed bioprosthetic valves. Eur Heart J. 2020 Aug 1;41(29):2731-2742. doi: 10.1093/eurheartj/ehaa544. PMID 32592401
- [Background] de Freitas Campos Guimaraes L, Urena M, Wijeysundera HC, Munoz-Garcia A, Serra V, Benitez LM, Auffret V, Cheema AN, Amat-Santos IJ, Fisher Q, Himbert D, Garcia Del Blanco B, Dager A, Le Breton H, Paradis JM, Dumont E, Pibarot P, Rodes-Cabau J. Long-Term Outcomes After Transcatheter Aortic Valve-in-Valve Replacement. Circ Cardiovasc Interv. 2018 Sep;11(9):e007038. doi: 10.1161/CIRCINTERVENTIONS.118.007038. PMID 30354588
- [Background] Wernly B, Zappe AK, Unbehaun A, Sinning JM, Jung C, Kim WK, Fichtlscherer S, Lichtenauer M, Hoppe UC, Alushi B, Beckhoff F, Wewetzer C, Franz M, Kretzschmar D, Navarese E, Landmesser U, Falk V, Lauten A. Transcatheter valve-in-valve implantation (VinV-TAVR) for failed surgical aortic bioprosthetic valves. Clin Res Cardiol. 2019 Jan;108(1):83-92. doi: 10.1007/s00392-018-1326-z. Epub 2018 Jul 12. PMID 30003366
- [Background] Webb JG, Murdoch DJ, Alu MC, Cheung A, Crowley A, Dvir D, Herrmann HC, Kodali SK, Leipsic J, Miller DC, Pibarot P, Suri RM, Wood D, Leon MB, Mack MJ. 3-Year Outcomes After Valve-in-Valve Transcatheter Aortic Valve Replacement for Degenerated Bioprostheses: The PARTNER 2 Registry. J Am Coll Cardiol. 2019 Jun 4;73(21):2647-2655. doi: 10.1016/j.jacc.2019.03.483. PMID 31146808
- [Background] Kaneko T, Makkar RR, Krishnaswami A, Hermiller J, Greenbaum A, Babaliaros V, Shah PB, Bailey SH, Bapat V, Kapadia S, Abbas AE. Valve-in-Surgical-Valve With SAPIEN 3 for Transcatheter Aortic Valve Replacement Based on Society of Thoracic Surgeons Predicted Risk of Mortality. Circ Cardiovasc Interv. 2021 May;14(5):e010288. doi: 10.1161/CIRCINTERVENTIONS.120.010288. Epub 2021 May 18. PMID 34003666
- [Background] Saxon JT, Allen KB, Cohen DJ, Chhatriwalla AK. Bioprosthetic Valve Fracture During Valve-in-valve TAVR: Bench to Bedside. Interv Cardiol. 2018 Jan;13(1):20-26. doi: 10.15420/icr.2017:29:1. PMID 29593832
- [Background] O'Donnell JP, O'Sullivan CJ. Bioprosthetic Aortic Valve Fracture During Valve-in-valve Transcatheter Aortic Valve Implantation. Interv Cardiol. 2019 Nov 18;14(3):147-151. doi: 10.15420/icr.2019.08.R2. eCollection 2019 Nov. PMID 31867060